CLINICAL TRIAL: NCT05672238
Title: Evaluation of Postoperative Acute Kidney Injury (AKI) Incidence and Risk Factors in Patients Underwent Pneumonectomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Bengi Safak (Unknown); Çiğdem Yıldırım Güçlü (Unknown); Basak Ceyda MECO (Unknown); Yusuf KAHYA (Unknown); Süleyman Gökalp Güneş (Unknown); İslam Aktürk (Unknown)
Responsible Party: Principal Investigator, Süheyla Karadağ Erkoç, Anesthesiology and Reanimation, Ankara University
Other Study IDs: AnkaraUPneumonectomyAKI
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury; Pneumonectomy; Status; Complication,Postoperative
Keywords: Acute Kidney Injury; Pneumonectomy
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a critical complication associated with a high incidence of morbidity and mortality that can occur in critically ill patients and after major surgical procedures. The aim of this study is to identify the incidance and outcomes of patients underwent pneumonectomy, defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a critical complication associated with a high incidence of morbidity and mortality that can occur in critically ill patients and after major surgical procedures. Although there is a decrease in pulmonary damage with restrictive fluid management and protective ventilatory strategies in patients who underwent wide lung resection to prevent pulmonary edema development after resection, the relative hypovolemia and hypoperfusion developed in patients may lead to renal dysfunction. The incidence of AKI after thoracic surgery can be up to 15% and is associated with prolonged length of stay (LOS) in hospital. The incidence of AKI is higher in patients with extensive resection such as pneumonectomy compared with lobectomy and wedge resection. Since AKI is not only a rare complication but also a risk factor for mortality, it is important to identify the incidence and risk factors of AKI, to prevent AKI and related complications and to improve patients outcomes. In this study incidence of AKI was defined using the KDIGO criteria according to the change of serum creatine levels.

166 patients who underwent pneumonectomy from January 2008 to December 2018 included the retrospective observational study. Demographic data, intraoperative data, rates of complications, risk factors for AKI, mortality, lenght of stay in intensive care unit (İCU) and hospital were evaluated. AKI was defined using the KDIGO criteria according to the serum creatinine levels. The SPSS 11.5 program was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent pneumonectomy, from January 2008 to December 2018

Exclusion Criteria:

* Chronic Kidney Disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent pneumonectomy
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury in patients underwent pneumonectomy | One week
  Kidney Disease Improving Global Outcomes (KDIGO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Karadağ Erkoç, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)